CLINICAL TRIAL: NCT05267834
Title: In Situ/Microinvasive Adenocarcinoma of the Uterine Cervix and HPV-type Impact: Pathologic Features, Treatment Options, and Follow-up Outcomes - Cervical Adenocarcinoma Study Group (CAS-Group).
Brief Title: Adenocarcinoma of the Uterine Cervix and HPV
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Luca Giannella, Principal Investigator, Università Politecnica delle Marche
Other Study IDs: AC-HPV2
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Adenocarcinoma of the Uterine Cervix
Keywords: Cervical Adenocarcinoma; HPV Type; Screening Program; Treatment; Recurrence; Survival; Follow-up
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive high-risk HPV: Women with adenocarcinoma of the uterine cervix and positive for high-risk HPV (genotype16/18/31/33/35/39/45/51/52/56/58/59/68).
  Interventions: Procedure: Conization and/or Hysterectomy
- Negative high-risk HPV: Women with adenocarcinoma of the uterine cervix and negative for high-risk HPV (genotype16/18/31/33/35/39/45/51/52/56/58/59/68).
  Interventions: Procedure: Conization and/or Hysterectomy

INTERVENTIONS:
Procedure: Conization and/or Hysterectomy — Women undergoing cervical conization or simple/modified/radical hysterectomy with or without pelvic lymphadenectomy

SUMMARY:
The present study will mainly aim to review and characterize the pathologic features, treatment options, and follow-up outcomes of women with in situ/microinvasive adenocarcinoma of the uterine cervix according to HPV status (positive versus negative high-risk HPV). It will evaluate the impact of HPV status on the recurrence and survival during a follow-up of five years. The present study will be a multi-institutional study including several oncological Italian Centers. Data will be retrospectively collected from January 2012 to December 2016 with a total follow-up of 5 years.

DETAILED DESCRIPTION:
The incidence of cervical cancer in developed countries declined considerably in the last few decades. This has been possible for efficient screening programs to which HPV vaccines have been added over the past 15 years. Despite this global reduction in cervical lesions, the incidence of adenocarcinoma of the uterine cervix (AC) increases in invasive and in situ stages. This increase mainly affects women aged 30-40, with an incidence of 11.2 per 100.000 women. On the contrary, the squamous histological lesions revealed an increase in the incidence of in situ lesions and a concomitant reduction of invasive stages. These data would seem to suggest a delay in the diagnosis of cervical glandular lesions, a shorter interval of disease progression from the adenocarcinoma in situ (AIS) to infiltrating stages, or a different process of carcinogenesis.

Most glandular cervical lesions occur at an early stage. The standard of treatment for in situ or micro-invasive lesions is extra fascial hysterectomy (AIS or stage 1A1 with no LVSI) or modified radical hysterectomy with pelvic lymph node dissection (stage 1A1 with LVSI, or 1A2). In fertility-sparing treatment, conization or radical trachelectomy with pelvic lymph node dissection is an option.

Another aspect that differentiates cervical adenocarcinoma from squamous lesions is the link with HPV infection. In 2018, the International Endocervical Criteria and Classification categorized cervical glandular lesions into HPV-associated and non-HPV-associated AC. Unlike cervical squamous lesions, which are almost all linked to high-risk HPV types, AC can be HPV negative in up to 15-20% of cases. The HPV 18 genotype is the most represented in AC with a rate of 38-50% in AIS and 50% in invasive stages. Based on some studies, it appears that non-HPV-related lesions have worse outcomes. This can significantly impact screening programs where 14 high-risk HPVs are tested.

In a recent study including 341 surgical specimens of AC, 100% of non-HPV-related lesions were classified as Silva Pattern C (the worst prognostic pattern). Instead, no impact of the HPV genotype was found on 113 women with AC during a follow-up of 5 years. HPV 45 showed a shorter 5-year survival than HPV 16 or 18.

While for advanced lesions, the stage itself represents the most important prognostic factor for prognosis, in situ or micro-invasive lesions may represent the best target for evaluating HPV status impact. This may be of interest as there is the option of conservative treatment in addition to standard treatment in early stages.

ELIGIBILITY:
Inclusion Criteria:

* Women with in-situ or microinvasive (stage 1A) adenocarcinoma of the uterine cervix undergoing conization or hysterectomy, between January 2012 and December 2016.
* Women with HPV testing within 2 months before conization.
* Women should be diagnosed and managed by the corresponding center.
* Patients with adequate clinical and pathological data.

Exclusion Criteria:

* Women with previous cervical treatments.
* Women with immunological disease (e.g. HIV).
* Unavailable HPV testing before surgery.
* Women with inadequate follow-up.

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women who were diagnosed with in situ or microinvasive (stage 1 A) adenocarcinoma of the uterine cervix, and undergoing surgical treatment, between 2012 and 2016.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Overall recurrence at 5 year in HPV positive vs HPV negative women | At 5 years
  Number of women who have recurrence after treatment divided by total number of patients at onset
Overall survival at 5 year in HPV positive vs HPV negative women | At 5 years
  Number of women who are alive after treatment divided by total number of patients at onset

SECONDARY OUTCOMES:
HPV-type disease recurrence at 5 years | At 5 years
  HPV genotypes associated with disease recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology and Obsetrics, Ancona, Italy

REFERENCES:
- [Result] Baalbergen A, Smedts F, Ewing P, Snijders PJ, Meijer CJ, Helmerhorst TJ. HPV-type has no impact on survival of patients with adenocarcinoma of the uterine cervix. Gynecol Oncol. 2013 Mar;128(3):530-4. doi: 10.1016/j.ygyno.2012.12.013. Epub 2012 Dec 19. PMID 23262207
- [Result] Liverani CA, Di Giuseppe J, Giannella L, Delli Carpini G, Ciavattini A. Cervical Cancer Screening Guidelines in the Postvaccination Era: Review of the Literature. J Oncol. 2020 Nov 5;2020:8887672. doi: 10.1155/2020/8887672. eCollection 2020. PMID 33204265
- [Result] Ciavattini A, Giannella L, De Vincenzo R, Di Giuseppe J, Papiccio M, Lukic A, Delli Carpini G, Perino A, Frega A, Sopracordevole F, Barbero M, Gultekin M. HPV Vaccination: The Position Paper of the Italian Society of Colposcopy and Cervico-Vaginal Pathology (SICPCV). Vaccines (Basel). 2020 Jul 2;8(3):354. doi: 10.3390/vaccines8030354. PMID 32630772
- [Result] Park KJ. Cervical adenocarcinoma: integration of HPV status, pattern of invasion, morphology and molecular markers into classification. Histopathology. 2020 Jan;76(1):112-127. doi: 10.1111/his.13995. PMID 31846527
- [Result] Fontham ETH, Wolf AMD, Church TR, Etzioni R, Flowers CR, Herzig A, Guerra CE, Oeffinger KC, Shih YT, Walter LC, Kim JJ, Andrews KS, DeSantis CE, Fedewa SA, Manassaram-Baptiste D, Saslow D, Wender RC, Smith RA. Cervical cancer screening for individuals at average risk: 2020 guideline update from the American Cancer Society. CA Cancer J Clin. 2020 Sep;70(5):321-346. doi: 10.3322/caac.21628. Epub 2020 Jul 30. PMID 32729638
- [Result] Talaat A, Brinkmann D, Dhundee J, Hana Y, Bevan J, Irvine R, Bailey S, Woolas R. Risk of significant gynaecological pathology in women with glandular neoplasia on cervical cytology. Cytopathology. 2012 Dec;23(6):371-7. doi: 10.1111/j.1365-2303.2011.00891.x. Epub 2011 Jul 12. PMID 21749501
- [Result] Koh WJ, Abu-Rustum NR, Bean S, Bradley K, Campos SM, Cho KR, Chon HS, Chu C, Clark R, Cohn D, Crispens MA, Damast S, Dorigo O, Eifel PJ, Fisher CM, Frederick P, Gaffney DK, Han E, Huh WK, Lurain JR, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Fader AN, Remmenga SW, Reynolds RK, Tillmanns T, Ueda S, Wyse E, Yashar CM, McMillian NR, Scavone JL. Cervical Cancer, Version 3.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Jan;17(1):64-84. doi: 10.6004/jnccn.2019.0001. PMID 30659131
- [Result] Teoh D, Musa F, Salani R, Huh W, Jimenez E. Diagnosis and Management of Adenocarcinoma in Situ: A Society of Gynecologic Oncology Evidence-Based Review and Recommendations. Obstet Gynecol. 2020 Apr;135(4):869-878. doi: 10.1097/AOG.0000000000003761. PMID 32168211
- [Result] Stolnicu S, Barsan I, Hoang L, Patel P, Terinte C, Pesci A, Aviel-Ronen S, Kiyokawa T, Alvarado-Cabrero I, Oliva E, Park KJ, Abu-Rustum NR, Pike MC, Soslow RA. Stromal invasion pattern identifies patients at lowest risk of lymph node metastasis in HPV-associated endocervical adenocarcinomas, but is irrelevant in adenocarcinomas unassociated with HPV. Gynecol Oncol. 2018 Jul;150(1):56-60. doi: 10.1016/j.ygyno.2018.04.570. Epub 2018 May 30. PMID 29859673
- [Result] Rositch AF, Soeters HM, Offutt-Powell TN, Wheeler BS, Taylor SM, Smith JS. The incidence of human papillomavirus infection following treatment for cervical neoplasia: a systematic review. Gynecol Oncol. 2014 Mar;132(3):767-79. doi: 10.1016/j.ygyno.2013.12.040. Epub 2014 Jan 7. PMID 24412508
- [Result] Perez S, Inarrea A, Perez-Tanoira R, Gil M, Lopez-Diez E, Valenzuela O, Porto M, Alberte-Lista L, Peteiro-Cancelo MA, Treinta A, Carballo R, Reboredo MC, Alvarez-Arguelles ME, Purrinos MJ. Fraction of high-grade cervical intraepithelial lesions attributable to genotypes targeted by a nonavalent HPV vaccine in Galicia, Spain. Virol J. 2017 Nov 6;14(1):214. doi: 10.1186/s12985-017-0879-1. PMID 29110680